CLINICAL TRIAL: NCT07209683
Title: Age-specific Neurovascular Effects of Transcranial Photobiomodulation
Brief Title: The Effect of Near-infrared Light Therapy on Brain Function and Cognition in Young and Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18356
Record Dates: First submitted 2025-09-26; First posted 2025-10-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cognition; Neurovascular Coupling Mechanism and Cognitive Function; Neurovascular Control; Brain Aging; Brain Activity
Keywords: transcranial photobiomodulation; neurovascular coupling; aging; cognitive function; near-infrared spectroscopy; electroencephalography; dynamic vessel analysis; home-based intervention; randomized double-blinded clinical trial

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group, double-blind, sham-controlled pilot trial. Healthy adult participants across multiple age groups (21-85 years) will be randomized in a 1:1 ratio to receive either active transcranial photobiomodulation (tPBM) or sham stimulation. Participants in both groups will complete 3-4 sessions per week for 4 weeks (20-minute sessions, every other day). Cognitive and physiological outcomes will be measured at baseline and post-intervention follow-up.
Who Masked: Participant, Outcomes Assessor
Masking Description: Unblinded and do not participate in outcome assessment and statistical analysis. These procedures are performed by blinded outcome assessors and blinded investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active near-infrared light therapy (Active Comparator): Participants in this arm will receive active transcranial photobiomodulation sessions every other day for 20 minutes during their participation in the study. The intervention will be administered by active Vielight Neuro Rx Gamma, a research version of a commercially available light therapy device categorized as a wellness product with non-significant risk. During these sessions, biologically effective near-infrared light will be administered.
  Interventions: Device: transcranial photobiomodulation
- Sham near-infrared light therapy (Sham Comparator): Participants in this arm will receive sham transcranial photobiomodulation sessions every other day for 20 minutes during their participation in the study. The intervention will be administered by active Vielight Neuro Rx Gamma, a research version of a commercially available light therapy device categorized as a wellness product with non-significant risk. During these sessions, biologically effective near-infrared light will not be administered.
  Interventions: Device: transcranial photobiomodulation

INTERVENTIONS:
Device: transcranial photobiomodulation — The Vielight Neuro Gamma TPBM devices (©Vielight Inc.) will be used to transmit pulsed near-infrared (NIR) energy through the cranium. Device emits NIR photons at 810 m wavelength generating ~100 mW/cm2 pulsed NIR power modulated at 40 Hz frequency. The six NIR light sources are positioned along the midline over the frontal, pariatel and occipital cortices, bilaterally over the temporal cortex, and intranasally. Due to its portable design, Vielight Neuro TBPM instruments can be used in the laboratory, bedside, or at the participant's home.
  Active / sham photobiomodulation sessions last for 20 minutes and will be administered at a laboratory-, home-, or office-based setting depending on the preference of the participant. TPBM will be performed three or four times a week for four weeks, maximum once every other day. Participants will complete a questionnaire of adverse events after each photobiomodulation session.
  Other Names: near-infrared light therapy

SUMMARY:
The goal of this pilot clinical trial is to test whether transcranial photobiomodulation (tPBM), a non-invasive brain stimulation technique using near-infrared light, can improve brain blood flow regulation (neurovascular coupling) and cognitive function in older adults.

The main questions it aims to answer are:

* Does tPBM enhance neurovascular coupling responses during memory and finger tapping tasks?
* Are these improvements linked to better cognitive performance and lower levels of brain inflammation and oxidative stress?

Researchers will compare an active tPBM treatment arm to a sham treatment arm to see if tPBM leads to measurable improvements in brain activity and cognitive function compared to no active stimulation.

Participants will:

* Receive either active tPBM or sham stimulation sessions for 4 weeks, every other day using a portable intervention device.
* Complete questionnaires and an iPAD-based cognitive testing protocol
* Complete memory and motor tasks while their brain activity is measured using non-invasive techniques: simultaneous functional near-infrared spectroscopy (fNIRS) and electroencephalography (EEG), transcranial doppler (TCD) flowmetry.
* Retinal vessel reactivity will be measured during flickering light stimulus using a special camera (dynamic vessel analysis, DVA).
* Provide blood samples to test for biomarkers of inflammation, oxidative stress and brain cell damage.

DETAILED DESCRIPTION:
Cognitive decline is a major cause of disability in older adults, and vascular pathologies play a critical role in the genesis of age-related cognitive impairment. Despite advances in understanding the pathophysiology of vascular cognitive impairment (VCI), effective interventions remain scarce. Neurovascular coupling (NVC), the physiological process that adjusts local cerebral blood flow to neuronal activity, is essential for maintaining optimal brain function. According to our preclinical and clinical studies, along with accumulating evidence from other research groups, dysregulation of NVC is increasingly recognized as a key contributor to age-related cognitive decline, highlighting an urgent need for targeted therapeutic strategies.

Transcranial photobiomodulation (tPBM) has emerged as a promising, non-invasive technique with the potential to enhance both neuronal and vascular health. tPBM delivers near-infrared light to cortical areas, stimulating mitochondrial activity, reducing oxidative stress, and improving cerebral hemodynamics. There is increasing evidence that tPBM, which uses red and infrared light with specific wavelengths, confers benefit in various neurological, cardiovascular, and cerebrovascular disorders. However, the underlying neurophysiological changes need to be clarified in human studies, and there are further patient populations who would benefit from a tPBM-based intervention. Optical imaging devices, such as near-infrared spectroscopy (NIRS), offer a means to evaluate tPBM-related changes in brain oxygenation and hemodynamics in an out-of-lab environment, which would significantly improve the feasibility of trials focusing on the effects of tPBM on cerebrovascular health. The practical advantages of tPBM lie in its documented safe application, simplicity of use, affordability, and the potential for home-based interventions.

Recent studies have demonstrated a strong association between cognitive performance and NVC responses in healthy older adults and in patients with mild cognitive impairment. Neuronal activity-induced vasodilation is largely mediated by nitric oxide (NO), whose dissociation from cytochrome c oxidase (CCO) and thus bioavailability is promoted by tPBM. It has also been shown that tPBM confers anti-inflammatory effects in the brain, which is relevant given the heightened inflammatory processes in older adult,s implicating aging-induced neuroinflammation. However, limited clinical evidence exists on the impact of tPBM on NVC, particularly in aging individuals. Moreover, existing research focuses on cognitive benefits rather than neurophysiological or hemodynamic changes, with minimal integration of these outcomes. Addressing this gap, this proposal aims to leverage advanced multimodal neuroimaging techniques to investigate the age-specific tPBM-improvements in NVC and its association with the effects on cognitive function.

Preclinical and early clinical studies suggest that tPBM enhances microvascular perfusion and tissue oxygenation, while simultaneously reducing neuroinflammation and oxidative stress. These dual effects underscore its potential as a multifaceted tool for promoting neural and vascular recovery. To date, evaluations of tPBM in various populations have shown it to be a safe intervention with transient and mild headache as the most common and considerable adverse effect induced by the sessions. Its non-pharmacological nature and compatibility with existing treatments further support its use as an innovative approach for cognitive rehabilitation.

The significance of this project lies in its potential to develop a novel, non-invasive intervention for cognitive impairment in aging populations and also in its ability to elucidate the underlying mechanisms of NVC modulation by tPBM. Findings from this research will provide critical insights into the dual neural and vascular effects of tPBM, laying the groundwork for future combination therapies to address age-related cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-85 years of age
* Adequate hearing and visual acuity to participate in the examinations
* Ability to read and write in English
* Competence to provide informed consent

Exclusion Criteria:

* Active CNS disease including multiple sclerosis, uncontrolled seizures, active brain cancer
* Cerebrovascular accident other than TIA within 60 days prior to Visit 0
* Major psychiatric disease, including major depression not currently controlled on medications, alcohol or drug abuse
* Participant currently uses commercial brain stimulation / neuromodulation device or an experimental device as part of a research study, e.g. tDCS, tACS, TBS, DBS, TMS, TPBM, etc.
* Participant currently takes dietary supplements with an expected cerebrovascular benefit, such as NAD- or NR-supplement, L-citrulline, urolithin
* Unstable medical condition, including uncontrolled diabetes, chronic heart issues, heart failure, chronic obstructive pulmonary disease, Stage 2 hypertension uncontrolled by medication (>160/100 mmHg)
* Any other medical condition or medication which, in the opinion of investigator, would render the patient inappropriate or too unstable to complete the study protocol.
* Pregnancy or trying to become pregnant in the next 1 months (self-reported), breastfeeding

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive performance | From baseline visit to the follow-up visit after completing a 4-week intervention protocol
  Cognitive performance will be assessed by using the following batteries of the NIH Toolbox: 1) Dimensional Change Card Sort [executive function]; 2) Pattern Comparison Processing Speed; 3) List Sorting Working Memory; 4) Flanker Inhibitory Control and Attention; 5) Picture Sequencing Memory and/or 6) Oral Symbol Digit Test.

SECONDARY OUTCOMES:
Neurovascular coupling response | From baseline visit to the follow-up visit after completing a 4-week intervention protocol
  Neuronal stimulus-induced cerebral hemodynamic response measured in the brain cortex using functional near-infrared spectroscopy, during a cognitive or motor paradigm. Increase in blood flow velocity recorded from the middle cerebral artery during cognitive n-back paradigm using transcranial Doppler (TCD) flowmetry.
Brain wave power | From baseline visit to the follow-up visit after completing a 4-week intervention protocol
  Band limited power in delta-, theta-, alpha-, beta- and gamma-bands during resting and task state measured by electroencephalography (EEG)
Functional connectivity | From baseline visit to the follow-up visit after completing a 4-week intervention protocol
  Correlation of simultaneously recorded cerebral hemodynamics (by fNIRS) or phase synchronization of simultaneously recorded cortical potential changes (by EEG).
Retinal vasoreactivity | From baseline visit to the follow-up visit after completing a 4-week intervention protocol
  Flickering light induced change in diameter of retinal arterioles and venules assessed by dynamic vessel analysis.

OTHER OUTCOMES:
Cerebrovascular endothelium-derived extracellular vesicles | From baseline visit to the follow-up visit after completing a 4-week intervention protocol
  Extracellular vesicles of cerebrovascular endothelial origin will be isolated from platelet poor plasma obtained from the participant and their count will be determined reflecting the health of brain vessels.
Pro-inflammatory cytokines | From baseline visit to the follow-up visit after completing a 4-week intervention protocol
  The following pro-inflammatory cytokines will be determined from participant's serum: Interleukin-1β, Interleukin-6, Interleukin-8 and Tumor Necrosis Factor-α

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Campus, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
IPD might not be shared due to the pilot nature of this clinical trial, which will be advertised locally.

REFERENCES:
- [Background] Chao LL. Effects of Home Photobiomodulation Treatments on Cognitive and Behavioral Function, Cerebral Perfusion, and Resting-State Functional Connectivity in Patients with Dementia: A Pilot Trial. Photobiomodul Photomed Laser Surg. 2019 Mar;37(3):133-141. doi: 10.1089/photob.2018.4555. Epub 2019 Feb 13. PMID 31050950